CLINICAL TRIAL: NCT01075438
Title: Descriptive Immunogenicity of 2 Doses of Pneumococcal 7-valent Conjugate Vaccine (Prevenar®, Wyeth Lederle) Followed by Pneumococcal Polysaccharide Vaccine (Pneumovax® Aventis Pasteur MSD) in Ataxia-telangiectasia Patients
Brief Title: Immunogenicity of Pneumococcal Vaccines in Ataxia-telangiectasia Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Galia Barkai, Sheba Medical Center
Other Study IDs: SHEBA-09-7444-GB-CTIL
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Ataxia Telangiectasia
Keywords: ataxia telangiectasia; Pneumococcal Vaccines
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for specific anti-pneumococcal antibody levels and Immunoglobulin levels.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Prevenar® (7-valent pneumococcal conjugate vaccine) — Pneumococcal vaccines (conjugate and polysaccharide)
  Intramuscular Injections: 2 doses of 7-valent pneumococcal conjugate vaccine 8 weeks apart and 1 dose of pneumococcal polysaccharide vaccine 8 weeks later
  Other Names: Prevenar®, Wyeth; Pneumovax® Aventis Pasteur MSD
Biological: Pneumovax® (pneumococcal polysaccharide vaccine) — Pneumococcal vaccines (conjugate and polysaccharide)
  Intramuscular Injections: 2 doses of 7-valent pneumococcal conjugate vaccine 8 weeks apart and 1 dose of pneumococcal polysaccharide vaccine 8 weeks later

SUMMARY:
Ataxia-telangiectasia (AT) is a rare genetic disorder characterized by gait disorders, neuromotor dysfunction, eye abnormalities and immune deficiency. AT patients are vulnerable to cancer and infection and usually die during their 2nd or 3rd decade due to these complications. The main cause of death is respiratory infections because these patients are known to have severe type of immunodeficiency. Consequently, pneumonia is the most common infection seen in AT patients, and is usually caused by S. pneumoniae. Therefore, a routine schedule of pneumococcal vaccine is highly recommended in AT cases where immunoglobulin replacement therapy was not already initiated.

Until recently, AT patients were immunized with the pneumococcal polysaccharide vaccine (PPV23, Pneumovax® Aventis Pasteur MSD). However, data have shown that they do not respond well to these vaccines. Recently, the Israeli Ministry of Health has approved the pneumococcal 7-valent conjugate vaccine (PCV7, Prevenar®, Wyeth Lederle) for AT patients of all ages. This conjugate vaccine is known to stimulate the immune system through a different mechanism and the response is expected to be higher. The approved Israeli schedule for immunization of AT patients includes children older than 2 years that are entitled to receive 2 doses of PCV7 (8 weeks apart) boosted by PPV23, eight weeks after the second dose of PCV7. Assessment of the antibody response of such pneumococcal vaccination protocol in AT patients has never been performed.

The "Safra" Children's Hospital is the national multi-disciplinary center caring for AT patients. Approximately 50 patients from all over the country (including Jewish, Druze, Bedouin and other Muslim patients - 3 of whom are Palestinians) are followed in the clinic on a monthly basis.

Approximately 20 AT patients are not receiving IVIG replacement therapy, therefore are entitled to receive pneumococcal vaccination as stated above (mean age 10.6, 3 -23 years, 3 less than 5 years)

The aim of this study is to evaluate the responsiveness, determined by specific antibody production, of AT patients receiving this new vaccine protocol.

DETAILED DESCRIPTION:
Ataxia-telangiectasia (AT) is a rare progressive neurodegenerative autosomal recessive disorder characterized by cerebellar ataxia, neuromotor dysfunction, oculocutaneous telangiectasia and immunodeficiency. AT patients are vulnerable to cancer and infection and usually die during their 2nd or 3rd decade due to these complications. Life expectancy does not correlate well with severity of neurological impairment. The main cause of death is respiratory infections because these patients are known to have severe type of immunodeficiency. The immunodeficiency of AT patient consists of both humoral defect (immunoglobulin deficiency and reduced response to polysaccharide antigens) and cell-mediated defect (reduced lymphocytes number and function). Consequently, pneumonia is the most common infection seen in AT patients, and is usually caused by S. pneumoniae. Therefore, a routine schedule of pneumococcal vaccine is highly recommended in AT cases where immunoglobulin replacement therapy was not already initiated.

Until recently, AT patients were immunized with the pneumococcal polysaccharide vaccine (PPV23, Pneumovax® Aventis Pasteur MSD). However, data have shown that they do not respond well to these vaccine mainly because of their reduced response to polysaccharide stimulation. Recently, the Israeli Ministry of Health has approved the pneumococcal 7-valent conjugate vaccine (PCV7, Prevenar®, Wyeth Lederle) for AT patients of all ages. In contrast to polysaccharide vaccines, this conjugate vaccine is known to stimulate the immune system through T-cell dependent mechanism, and therefore the response is expected to be higher. The approved Israeli schedule for immunization of AT patients includes children older than 2 years that are entitled to receive 2 doses of PCV7 (8 weeks apart) boosted by PPV23, eight weeks after the second dose of PCV7. Assessment of the immunogenicity of such pneumococcal vaccination protocol in AT patients has never been performed.

The "Safra" Children's Hospital is the national multi-disciplinary center caring for AT patients. Approximately 50 patients from all over the country (including Jewish, Druze, Bedouin and other Muslim patients - 3 of whom are Palestinians) are followed in the clinic on a monthly basis.

Approximately 20 AT patients are not receiving IVIG replacement therapy, therefore are entitled to receive pneumococcal vaccination as stated above (mean age 10.6, 3 -23 years, 3 less than 5 years.

The aim of this study is to evaluate the responsiveness, determined by specific antibody production, of AT patients receiving the new vaccine protocol that was recently approved to use by the Israeli Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

1. AT patients attending the national AT clinic
2. 2+ years of age
3. Agree to join this study

Exclusion Criteria:

1. Patients on regular immunoglobulin replacement therapy (other patients who are not on replacement therapy but have received IVIG 3 months or less before the beginning of the study)
2. Current infection
3. Previous serious adverse reactions to vaccination
4. Administration of other vaccines within 4 weeks before administration of study vaccine or plan for vaccination 26 weeks following the first vaccine (PCV7)

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ataxia Telangiectasia patients, not cuurntly on replacement Immunoglobulin G therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Primary end point will be levels of antibodies against 13 serotypes of streptococcus pneumoniae following vaccination with 2 doses of PCV7 and 1 dose of PPV23. All endpoints will include both ELISA and OPA antibodies. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel